CLINICAL TRIAL: NCT04346160
Title: Tear Fluid miRNA Analysis in Sars-Cov2 Conjunctivitis
Brief Title: A Study to Assess the Virus RNA, and miRNA Levels Related to Viral Infection, and Inflammatory Response in Tears of Patients Affected by COVID-19 Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Leonardo Mastropasqua, Study Director, Professor, G. d'Annunzio University
Other Study IDs: UChieti03
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: COVID; Conjunctivitis
Keywords: COVID; conjunctivitis; SARS-CoV2; miRNA; tear fluid
MeSH Terms: conditions — Conjunctivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tear fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with bilateral conjunctivitis: Hospitalized patient affected by COVID-19 disease with bilateral conjunctivitis defined as red eyes (macroscopic signs of conjunctival congestion)
  Interventions: Diagnostic Test: Schirmer Test I
- Patients without conjunctivitis: Hospitalized patient affected by COVID-19 disease without any signs of conjunctivitis defined as red eyes (macroscopic signs of conjunctival congestion)
  Interventions: Diagnostic Test: Schirmer Test I
- Healthy control group: group of healthy patients considered as controls
  Interventions: Diagnostic Test: Schirmer Test I

INTERVENTIONS:
Diagnostic Test: Schirmer Test I — Collection of tear fluid

SUMMARY:
The aim of this study is to assess the virus RNA, and miRNA levels related to viral infection, and inflammatory response in tears of hospitalized patients with a diagnosis of COVID-19 with and without conjunctivitis and to correlate them with clinical condition.

Tears will be collected by using Schirmer Test I, a non invasive painless test which can be performed at the patient's bed. Tears will be collected on the graduated paper strips pulling the lower lid gently downward for 5 minutes. Following, the strip will be placed in a 2.0 mL Eppendorf tube and stored at -80◦C (or - 20°C)

DETAILED DESCRIPTION:
The SARS-CoV-2 is a virus highly infectious whose main target of infection is the respiratory tract. Virus has been reported to target other mucus tissues, such as the conjunctiva of the eye and causes conjunctivitis. A recent study has detected the presence of SARS-CoV-2 in the tears of patients affected by COVID-19 with conjunctivitis, using real-time reverse transcription polymerase chain reaction (RT-PCR). This suggests that droplets and body fluids of infected people can contaminate the human conjunctival mucosa and it can be a view of transmission that it must not be ignored.

A role of miRNAs has been found in ocular infections such as fungal, bacterial, viral infections. It would be interesting to correlate tear fluid miRNA levels to patients clinical findings

ELIGIBILITY:
Inclusion Criteria (Group 1):

* A confirmed diagnosis of COVID-19 disease
* Age ≥ of 18 years.
* absence of conjuntivitis detected by portable slit lamp

Inclusion Criteria (Group 2):

* A confirmed diagnosis of COVID-19 disease
* Age ≥ of 18 years.
* Presence of bilateral conjunctivitis defined as red eyes (macroscopic signs of conjunctival congestion)

Exclusion Criteria (both groups):

* Pregnant women
* Any form Ocular surface diseases preceding Covid-19 diagnosis, Glaucoma, history of anterior segment inflammation, previous penetrating ocular trauma
* Ocular surgeries within previous 6 months
* Topical therapies
* History of ocular allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a total of 25 patients with a diagnosis of COVID-19 with bilateral conjunctivitis (Group 1) and without conjunctivitis (Group 2) will be enrolled at the Anesthesia and Intensive Care department, the Infectious diseases department and the Emergency Medicine department, at the "SS. Annunziata Hospital" of Chieti-University G. D'Annunzio, Chieti-Pescara, Italy, in April 2020. A group of healthy patients will be enrolled and were considered as controls
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-04-14 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
virus molecular analysis | 2 weeks
  - to asses virus RNA and miRNA levels in tears
host molecular analysis | 2 weeks
  - to asses inflammatory response molecules

SECONDARY OUTCOMES:
Epidemiologic data | 2 weeks
  To analyze the prevalence of conjunctivitis in patients with a diagnosis of COVID-19 and the assessment of the predictive value of conjunctivitis in the development of the COVID-19 disease (or in developing respiratory distress forms-ARDS).

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Mastropasqua, Professor, Principal Investigator — Ophtalmology Clinic, G. d'Annunzio University
Locations (1):
- Ophtalmology Clinic, G.d'Annunzio University, Chieti, Italy